CLINICAL TRIAL: NCT03716102
Title: OPTIMIZE Sirolimus-Eluting Coronary Stent Systems Pharmacokinetics (PK) Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Svelte Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IP-18-001
Record Dates: First submitted 2018-10-18; First posted 2018-10-23 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Svelte DES (Experimental): Stent: A mounted Cobalt Chromium (Co-Cr) alloy based stent Polymer coating: Polyesteramide (PEA) Sirolimus drug
  Interventions: Device: PCI with implantation with DES

INTERVENTIONS:
Device: PCI with implantation with DES — PCI with implantation with DES

SUMMARY:
To evaluate the pharmacokinetic parameters of sirolimus release from the Svelte DES.

DETAILED DESCRIPTION:
This is a prospective, open, non-randomized, study involving two (2) centers in the United States. A minimum of twelve (12) and a maximum of fifteen (15) subjects will be consented, treated and have blood samples drawn to evaluate the pharmacokinetic parameters of sirolimus release from the Svelte DES.

ELIGIBILITY:
Inclusion Criteria:

* Subject is an eligible candidate for PCI
* Subject has symptomatic coronary artery disease with objective evidence of ischemia or silent ischemia
* Subject is an acceptable candidate for CABG
* Subject has ≤ 3 de novo target lesions in ≤ 2 native coronary artery vessels, with ≤ 2 lesions in a single vessel, each meeting the angiographic criteria and none of the exclusion criteria
* Target lesion(s) must be located in a native coronary artery with RVD ≥ 2.25mm and ≤ 4.00mm

Exclusion Criteria:

* Subject has cardiogenic shock, hemodynamic instability requiring inotropic or mechanical circulatory support, intractable ventricular arrhythmia, or ongoing intractable angina
* Subject's target lesion(s) is located in the left main coronary artery
* Subject's target lesion(s) is located within 3mm of the origin of the LAD or LCX coronary artery
* Subject's target lesion(s) is located within a SVG or an arterial graft
* Subject's target lesion(s) will be accessed via SVG or arterial graft

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2018-11-21 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2021-07-15 (Estimated)

PRIMARY OUTCOMES:
Maximum observed blood concentration (Cmax) | Up to 30 days
Time to reach maximum blood concentration (tmax) | Up to 30 days
Area under the blood concentration versus time curve: time zero to the final quantifiable concentration) (AUC 0-t) | Up to 30 days
Area under the blood concentration versus time curve: time zero to the extrapolated infinite time (AUC 0-∞) | Up to 30 days
Terminal phase half-life (t1/2) | Up to 30 days
Apparent total blood clearance (CL/F) | Up to 30 days
Apparent volume of distribution (Vd/F) | Up to 30 days

SECONDARY OUTCOMES:
Target Vessel Failure (TVF) | 6 months, 12 months, 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Donohoe, MD, Study Director — Svelte Medical Systems
Locations (2):
- United States (2):
  - Scottsdale Healthcare, Scottsdale, Arizona
  - Northern Michigan Hospital d.b.a McLaren Northern Michigan, Petoskey, Michigan

IPD SHARING:
Plan to Share IPD: No